CLINICAL TRIAL: NCT05480215
Title: Prospective Study for Symptomatic Relief of Action Tremor With Cala Trio Using Trio+ Bands
Brief Title: Symptomatic Relief of Action Tremor With Cala Trio Using Trio+ Bands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cala Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ET-22
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Essential Tremor; Parkinson Disease
MeSH Terms: conditions — Essential Tremor; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental: TAPS delivered by Cala device with Trio band (Experimental): Two 40-minute TAPS sessions daily for 14 days
  Interventions: Device: Cala Device
- Experimental: TAPS delivered by Cala device with Trio+ band (Experimental): Two 40-minute TAPS sessions daily for 14 days
  Interventions: Device: Cala Device

INTERVENTIONS:
Device: Cala Device — transcutaneous afferent patterned stimulation (TAPS)

SUMMARY:
Demonstrate safety and effectiveness of symptomatic action tremor relief in the treated hand following stimulation with the Cala Trio System using the Trio+ bands as compared to the Trio bands in adults with Essential Tremor (ET) and/or Parkinson's Disease (PD) over 2 weeks.

DETAILED DESCRIPTION:
20 patients with (13 with ET and 7 with PD) with at least mild postural tremor were enrolled in a prospective, single-center, two-arm, crossover study that took place over the course of four weeks. TAPS devices were shipped to patients to run the study remotely. In the first arm of the study, subjects received TAPS treatment using the original. Cala Trio band for two weeks. Followed by a wash-out period (> 24 hours), subjects entered the second arm and received TAPS using the Trio+ band for an additional two weeks. Unsupervised motion assessments were captured at home, and at the beginning and end of the four weeks by telemedicine.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥22 years of age
* Competent and willing to provide written, informed consent to participate in the study
* Willing to comply with study protocol requirements

For subjects with Essential Tremor:

* A diagnosis of essential tremor
* A tremor severity score of 2 or above in the dominant hand/arm as measured by one of the TETRAS upper limb postural tremor items
* No significant alcohol intake within 8 hours prior to study visits

For subjects with Parkinson's Disease:

* Dominant hand/arm exhibiting postural tremor ≥ 2 (while in the off state) as assessed by the MDS-UPDRS postural tremor score
* Stable dose of Parkinson's disease medications, if applicable, for 30 days prior to study entry

Exclusion Criteria:

* Implanted electrical medical device, such as a pacemaker, defibrillator, or deep brain stimulator
* Suspected or diagnosed epilepsy or other seizure disorder
* Any skin condition at the stimulation site that in the investigator's opinion should preclude participation in this study
* Diagnosed with peripheral neuropathy affecting the tested upper extremity
* Presence of any other neurodegenerative disease other than essential tremor or Parkinson's Disease
* Subjects unable to communicate with the investigator and staff
* Any health condition or concomitant medication that in the investigator's opinion should preclude participation in this study
* Pregnancy or anticipated pregnancy during the course of the study
* Botulinum toxin injection for hand tremor within 6 months prior to study enrollment
* Are participating or have participated in another interventional clinical trial in the last 30 days which may confound the results of this study, unless approved by the Sponsor

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Tremor power changes from pre-stimulation to post-stimulation | baseline, pre-intervention and immediately after the intervention
  Tremor improvement was measured by Tremor Power Improvement Ratio (TPIR) using kinematic data collected by the device. The TPIR was calculated as pre-stimulation power divided by post-stimulation power, which was computed from device-collected accelerometer data

SECONDARY OUTCOMES:
Change in TETRAS from pre-stimulation to post- stimulation within each visit | baseline, pre-intervention and immediately after the intervention
  For subjects with Essential Tremor only: Tremor Research Group Essential Tremor Rating Assessment Scale (TETRAS) subset score, relevant to the stimulated upper limb, change from pre-stimulation to post- stimulation within each visit
Change in UPDRS Part III from pre-stimulation to post- stimulation within each visit | baseline, pre-intervention and immediately after the intervention
  For subjects with Parkinson's Disease only: Modified Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS) subset score, change from pre- stimulation to post-stimulation within each visit
Change in BF-ADL | baseline, pre-intervention and immediately after the intervention
  Change in the Bain & Findley activities of daily living (BF-ADL) score from pre- to post-stimulation at each of the two study visits associated with the Trio and Trio+ bands (four study visits total)

CONTACTS AND LOCATIONS:
Locations (1):
- Cala Clinic, San Mateo, California, United States